CLINICAL TRIAL: NCT07176728
Title: A Single-blind, Placebo Controlled, Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BAY 3389934 Intravenous Infusions in Healthy Japanese Participants.
Brief Title: A Study to Assess the Safety and Effects of Different Doses of an Investigational Drug, BAY 3389934, in Healthy Japanese Volunteers.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 22371
Record Dates: First submitted 2025-08-29; First posted 2025-09-16 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Sepsis Associated Disseminated Intravascular Coagulation (DIC)
Keywords: Sepsis, Disseminated Intravascular Coagulation, Coagulopathy
MeSH Terms: conditions — Sepsis; Disseminated Intravascular Coagulation; Hemostatic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Step 1 BAY 3389934 (Experimental): 15 mg/h/ intravenous Single Dose for 4 h fasting
  Interventions: Drug: BAY 3389934
- Dose Step 2 BAY 3389934 (Experimental): Max. dose 35 mg / h / intravenous - actual dose will be determined after Dose Step 1 Single Dose for 4 h fasting
  Interventions: Drug: BAY 3389934
- Dose Step 1 and Dose Step 2 Placebo (Placebo Comparator): Placebo / intravenous Single Dose for 4 h Fasting
  Interventions: Drug: Matching Placebo / Diluent

INTERVENTIONS:
Drug: BAY 3389934 — Solution for intravenous infusion
  Arms: Dose Step 1 BAY 3389934; Dose Step 2 BAY 3389934
Drug: Matching Placebo / Diluent — Solution for intravenous infusion
  Arms: Dose Step 1 and Dose Step 2 Placebo

SUMMARY:
This study is designed to evaluate a new investigational drug, BAY 3389934, in healthy Japanese volunteers. The primary purpose is to see how safe the drug is and how well it is tolerated by the body when given at different doses. BAY 3389934 is being developed for the potential treatment of a serious blood clotting condition called sepsis-associated disseminated intravascular coagulation (DIC). The research will be conducted as a single-blind, placebo-controlled, dose-escalation study. This means that participants will be randomly assigned to receive either the active drug (BAY 3389934) or a placebo (an inactive substance), and they will not know which one they are receiving. The study will involve up to 16 healthy male and female Japanese participants, aged between 18 and 55. The study consists of two parts, called dose steps. In the first step, participants will receive a single 4-hour intravenous (IV) infusion of BAY 3389934 at a dose of 15 mg/h, or a placebo. Based on the safety and tolerability results from this first step, a second, higher dose will be selected for the next group of participants in the second step. Throughout the study, researchers will closely monitor participants for any side effects (adverse events). They will also collect blood and urine samples to study how the drug is absorbed, distributed, and eliminated by the body (pharmacokinetics or PK) and what effects it has on the body's clotting system (pharmacodynamics or PD). This involves measuring specific substances in the blood, such as activated partial thromboplastin time (aPTT) and prothrombin time (PT). Participants will stay at the study center for 4 days and will have a follow-up visit 3 to 5 days after they are discharged. The information gathered from this study is crucial for the future clinical development of BAY 3389934 in Japan and for designing future studies in patients with septic DIC.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive.

  * Participants who are overtly healthy Japanese as determined by medical evaluation.
  * Body mass index (BMI) within the range 18 - 29.9 kg/m² (inclusive).
  * Male participants must agree to use specified contraception during the study and for at least 90 days plus 5 half-lives after.
  * Female participants must be a Woman of Nonchildbearing Potential (WONCBP).
  * Capable of giving signed informed consent.
  * Willing to comply with the requirements and restrictions listed in the protocol.

Exclusion Criteria:

* Any medical disorder, condition, or history that would impair participation.

  * Known hypersensitivity to the study drug or its excipients.
  * Known disorders with increased bleeding risk or known congenital/acquired coagulation disorders.
  * Use of prescription drugs, over-the-counter drugs, or herbal products within 14 days or 5 half-lives before the study.
  * Clinically relevant findings in the ECG, such as a QTcF over 450 msec.
  * Systolic blood pressure below 90 mmHg or above 140 mmHg at screening and admission.
  * Diastolic blood pressure below 40 mmHg or above 90 mmHg at screening and admission.
  * Positive results for Hepatitis B, Hepatitis C, or HIV.
  * Positive drug screening, alcohol breath test, or urine cotinine test.
  * Clinically relevant deviations of the screened laboratory parameters from reference ranges at the screening visit.
  * Positive pregnancy test.
  * Donation of blood or plasma within specified timeframes before the study.
  * Lack of compliance with lifestyle restrictions (e.g., alcohol, specific foods, strenuous activity).
  * Previous participation in this or another clinical study within a specified timeframe.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From start of study intervention until the follow-up visit (approximately 5 weeks)
  Investigate the safety and tolerability of BAY 3389934 15 mg/h and a second, higher dose (will be determined based on the result of 15 mg/h dose step), 4-hours infusion, respectively.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Profile of BAY 3389934 - Cmax | From pre-dose (0 hours) up to 48 hours after start of infusion
  Maximum observed drug concentration (Cmax) within the given timeframe. PK parameters will be calculated using the non-compartmental method according to the sponsor's current guidelines using PhoenixTM (Certara, Princeton, New Jersey).
Pharmacokinetic (PK) Profile of BAY 3389934 - AUC | From pre-dose (0 hours) up to 48 hours after start of infusion
  Area under the concentration vs. time curve from zero to infinity (AUC) within the given timeframe. In the case of an unexpected event of e.g., an exceedingly large (>20%) extrapolated portion of AUC (AUC(tlast-∞)), the parameter AUC(0-tlast) may be evaluated as main parameter. PK parameters will be calculated using the non-compartmental method according to the sponsor's current guidelines using PhoenixTM (Certara, Princeton, New Jersey).
Pharmacokinetic (PK) Profile of BAY 3389934 - Cmax/D | From pre-dose (0 hours) up to 48 hours after start of infusion
  Maximum observed drug concentration (Cmax) divided by dose (Cmax/D) within the given timeframe. PK parameters will be calculated using the non-compartmental method according to the sponsor's current guidelines using PhoenixTM (Certara, Princeton, New Jersey).
Pharmacokinetic (PK) Profile of BAY 3389934 - AUC/D | From pre-dose (0 hours) up to 48 hours after start of infusion
  Area under the concentration vs. time curve from zero to infinity (AUC) divided by dose (AUC/D) in the given timeframe. In the case of an unexpected event of e.g., an exceedingly large (>20%) extrapolated portion of AUC (AUC(tlast-∞)), the parameter AUC(0-tlast) may be evaluated as main parameter. PK parameters will be calculated using the non-compartmental method according to the sponsor's current guidelines using PhoenixTM (Certara, Princeton, New Jersey).
Pharmacokinetic (PK) Profile of BAY 3389934 - t 1/2 | From pre-dose (0 hours) up to 48 hours after start of infusion
  Half-life associated with the terminal slope (t1/2) of BAY 3389934 in plasma within the given timeframe.
  PK parameters will be calculated using the non-compartmental method according to the sponsor's current guidelines using PhoenixTM (Certara, Princeton, New Jersey).
Pharmacodynamic (PD) Profile of BAY 3389934 - aPTT | From pre-dose up to 5 hours after beginning of infusion.
  Measure Activated partial thromboplastin time (aPTT). Assessed as the maximal ratio to baseline and the ratio to baseline at 4 hours and 5 hours after beginning of infusion.
Pharmacodynamic (PD) Profile of BAY 3389934 - PT | From pre-dose up to 5 hours after beginning of infusion.
  Prothrombin time (PT). Assessed as the maximal ratio to baseline and the ratio to baseline at 4 hours and 5 hours after beginning of infusion.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - SOUSEIKAI Fukuoka Mirai Hospital, Fukuoka, Fukuoka Pref
  - SOUSEIKAI Fukuoka Mirai Hospital, Fukuoka

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.